CLINICAL TRIAL: NCT00999310
Title: Neuropsychologic, Neuroradiologic, Endocrinologic, and Genetic Aspects of Klinefelter Syndrome
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M-20080238
Record Dates: First submitted 2009-10-20; First posted 2009-10-21 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2012-09

CONDITIONS: Klinefelter Syndrome
Keywords: Klinefelter syndrome; Neuropsychology; Neuroradiology; Genetics
MeSH Terms: conditions — Klinefelter Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Klinefelter syndrome
- Control men
- Control women
- parents of Klinefelter groupe

SUMMARY:
The purpose of this study is to investigate the following:

1. Whether Klinefelter Syndrome is associated with altered total and regional brain volumes and altered brain activity.
2. The influence of genetic factors and testosterone treatment on the neuropsychological phenotype, total and regional brain volumes and brain activity in men with Klinefelter syndrome.

DETAILED DESCRIPTION:
Klinefelter syndrome (KS) is the most common sex-chromosome disorder in men with a prevalence of 1 in 660 men. Men with the syndrome have an additional X-chromosome. The syndrome is associated with cognitive and behavioral dysfunction and also with hypogonadism. Magnetic resonance imaging have pointed to different volumetric alterations in several brain structures. Several genetic factors involving the X-chromosome have been suggested to influence the neuropsychological phenotype in men with KS.

The aim of this study is to investigate the following: 1.Whether KS is associated with altered total and regional brain volumes and altered brain activity. 2.Whether genetic factors influence the neuropsychological phenotype, total and regional brain volumes, and brain activity in men with KS. 3.Whether testosterone treatment improves cognitive skills and change brain activity in men with KS.

Participants are divided in 5 groups: 1. 50 men with KS who receive testosterone treatment. 2. 50 men KS who do not receive testosterone treatment. 3. 100 age-matched control men.4. 50 age-matched control women are included as a control group for X-chromosome inactivation pattern. 5. Parents of KS subjects in group 1 and 2 are included to determine the parental origin of the supernumerary X-chromosome. Methods include a 3-hour battery of standardized neuropsychological tests to cover a broad range of cognitive domains and to assess major domains of personality. We use magnetic resonance imaging to measure total and regional brain volumes and functional magnetic resonance imaging to measure brain activity while subjects are performing a attention-demanding cognitive task. The genetic testing includes the parental origin of the supernumerary X-chromosome, the pattern of X-chromosome inactivation, androgen receptor (AR) CAGn repeat length, and gene expression profile of brain-expressed genes.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 60 years
* verified KS karyotype (KS patients)

Exclusion Criteria:

* present or past neurological diseases
* present or past head trauma
* contraindication to perform MR scans(Claustrophobia,Magnetic or electric foreign bodies - including cardiac pacemakers, magnetic cerebrovascular clips and electric non-removable appliances dosing medicine)
* extreme adiposity (BMI > 35 kg/m2)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Klinefelter syndrome are recruited from endocrine and fertility clinics.
  The control groups are recruited by advertising for healthy volunteers at the University of Aarhus and at the Blood Bank at the Aarhus University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claus H Gravholt, MD, DMSCI, Principal Investigator — Medical Department M, Endocrinology and Diabetes, and Medical Research Laboratories, Clinical Institute, Aarhus University Hospital, Aarhus, Denmark; Anne S Jensen, MD, Principal Investigator — University of Aarhus
Locations (1):
- Medical Department M, Endocrinology and Diabetes, and Medical Research Laboratories, Clinical Institute, Aarhus University Hospital, Nørrebrogade 44, Aarhus, Denmark

REFERENCES:
- [Derived] Viuff M, Skakkebaek A, Johannsen EB, Chang S, Pedersen SB, Lauritsen KM, Pedersen MGB, Trolle C, Just J, Gravholt CH. X chromosome dosage and the genetic impact across human tissues. Genome Med. 2023 Mar 28;15(1):21. doi: 10.1186/s13073-023-01169-4. PMID 36978128
- [Derived] Chang S, Skakkebaek A, Trolle C, Bojesen A, Hertz JM, Cohen A, Hougaard DM, Wallentin M, Pedersen AD, Ostergaard JR, Gravholt CH. Anthropometry in Klinefelter syndrome--multifactorial influences due to CAG length, testosterone treatment and possibly intrauterine hypogonadism. J Clin Endocrinol Metab. 2015 Mar;100(3):E508-17. doi: 10.1210/jc.2014-2834. Epub 2014 Dec 16. PMID 25514102
- [Derived] Skakkebaek A, Bojesen A, Kristensen MK, Cohen A, Hougaard DM, Hertz JM, Fedder J, Laurberg P, Wallentin M, Ostergaard JR, Pedersen AD, Gravholt CH. Neuropsychology and brain morphology in Klinefelter syndrome - the impact of genetics. Andrology. 2014 Jul;2(4):632-40. doi: 10.1111/j.2047-2927.2014.00229.x. Epub 2014 May 28. PMID 24865607